CLINICAL TRIAL: NCT03633214
Title: Evaluation of An Online Intervention In Improving General Practitioners' Practice In Prostate Cancer Screening
Acronym: ProCaSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Tun Firzara Abdul Malik, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BK070-2016
Record Dates: First submitted 2018-08-01; First posted 2018-08-16 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer Screening
Keywords: Prostatic neoplasms; Mass screening; General practitioners; Primary health care; Clinical trial
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training module (Intervention) (Active Comparator): Responses of GPs in the intervention group will then be compared before and immediately after the online training video and also 3-months later
  Interventions: Other: Online training module
- No training module (Control) (No Intervention)

INTERVENTIONS:
Other: Online training module — Responses of GPs in the intervention group will then be compared before and immediately after the online training video and also 3-months later; as well as to the control group.
  Arms: Training module (Intervention)

SUMMARY:
The incidence of prostate cancer has been rising steadily both globally and in Malaysia. Besides an ageing population, another reason cited to explain the increase, is the corresponding increase in the prostate cancer screening rates, especially using non-invasive tests like the prostate specific antigen (PSA).

General practitioners, being front liners in medicine, play an important role in helping men make an informed decision on prostate cancer screening. In Malaysia, about 50% of GPs would routinely screen asymptomatic men and 95% of them would use PSA as a screening tool. Despite this, the evidence for screening is inconclusive, as evidenced from two major trials on screening [The European Randomised Study of Screening for Prostate Cancer (ERSPC) and Prostate, Lung, Colorectal and Ovarian Cancer Screening trial (PLCO)]. Furthermore, clinical practice guidelines globally provide conflicting recommendations on this subject, and none has been published in Malaysia to date.

Therefore, our study aims to determine the effectiveness of an online training module in helping GPs' better understand the controversies surrounding prostate cancer screening, and in so doing, improve their practice of screening. The investigators hypothesise that GPs who are randomised to receive their online module will be less inclined to screen unnecessarily for prostate cancer.

DETAILED DESCRIPTION:
Study design: Randomised controlled trial

Setting: This trial will involve GPs in the Klang Valley, encompassing the Petaling district and Kuala Lumpur.

The healthcare system in Malaysia is divided into public and private sectors. Patients pay a standard minimal fee for public healthcare system whereas the private sector charges patients based on the services provided. The study will be conducted in private GP clinics as PSA testing is readily available compared to the public primary care setting. In public primary care clinics, PSA screening is not offered as part of a routine screening programme.

Sample size:

With 80% power and 5% (two-sided) significance, with an estimated 40% reduction in PSA screening from baseline in the intervention group and 10% in the control group, the number of participants needed for each group is 38 (total 76). Therefore, a total of 96 GPs in the Klang Valley will be recruited for this study, assuming a non-response rate of 20 GPs.

Intervention:

The intervention consists of two phases.

Phase 1 The research team will develop 3 self-administered, online surveys, with the input of family physicians and urologists. The surveys will capture basic demographic information about the participating GPs (but not any identifiable information), and also their overall knowledge and perception towards prostate cancer screening. In addition, all 3 surveys will also contain 5 clinical vignettes that will relate to prostate cancer screening. After reading the vignettes, the GPs will be asked whether or not they would recommend screening for the particular patient in the given scenario; and should they choose to screen, which screening method they would use (PSA, DRE, or both).

GPs will then be randomised to either receive an online training module (intervention) or none (control).

Phase 2:

Upon successful receipt of the GPs' response to the first survey, a second survey will be sent to all the GPs via email. The participants will once again be invited to read and respond to another set of vignettes of similar nature to those in phase 1.

GPs who have been randomised to the intervention arm will also receive a link in the second email that will enable them to download an online training module. The participants will be asked to view the training module prior to answering the second survey.

GPs in the control group will only receive the second survey and not the training module.

A third and final email will be sent to all the GPs who have successfully answered the second survey, 3 months after the date of receipt of their second survey response. This final survey will likewise, contain five clinical vignettes of similar nature to those of the two previous surveys. The responses of GPs in the intervention group will then be compared before and immediately after the online training video and also 3-months later; as well as to the control group.

Recruitment:

The research team will recruit the GPs from an existing GP database which has been created from previous studies conducted in the Petaling District and Kuala Lumpur. A researcher and a research assistant will be responsible for identifying and recruiting eligible participants. An invitation letter, a study summary, a participant information sheet and consent form will be sent via email to each GP. Consenting participants will be remunerated for their time and effort spent in participating in the study. In the event response is poor, a research assistant may need to arrange an appointment to visit the GPs at their clinics'.

Analysis:

The McNemar test will be used to determine the phase differences in the proportion of GPs who perform screening unnecessarily and the differences between the intervention and control group. Chi square test will be used to compare the difference in proportions between the intervention and control groups. GPs' characteristics associated with unnecessary screening practice will be explored using logistic regression models using phase 1 data. Logistic regression will be used for binary outcomes and the analyses will be adjusted for baseline data. SPSS will be used to manage the data sets

ELIGIBILITY:
Inclusion Criteria:

* Full time general practitioners in the Klang valley (Petaling district and Kuala Lumpur)

Exclusion Criteria:

* GPs who do not see male patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of effectiveness of online training module among general practitioners in prostate cancer screening | Through study completion, an average of 6 months
  Difference in the change in proportions of appropriate prostate cancer screening from baseline by GPs between intervention (online training module) and control (no online training module) groups.

SECONDARY OUTCOMES:
Post-online training module knowledge in prostate cancer screening | An average of 6 months
  1. Difference in the post-online training module knowledge and attitudes towards prostate cancer screening between the intervention and control groups.
  2. GPs' characteristics that are associated with prostate cancer screening

CONTACTS AND LOCATIONS:
Overall Officials: Tun Firzara Abdul Malik, Principal Investigator — University of Malaya
Locations (1):
- Department of Primary Care Medicine, University of Malaya Medical Centre, Kuala Lumpur, Lembah Pantai, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Ciatto S, Nelen V, Kwiatkowski M, Lujan M, Lilja H, Zappa M, Denis LJ, Recker F, Paez A, Maattanen L, Bangma CH, Aus G, Carlsson S, Villers A, Rebillard X, van der Kwast T, Kujala PM, Blijenberg BG, Stenman UH, Huber A, Taari K, Hakama M, Moss SM, de Koning HJ, Auvinen A; ERSPC Investigators. Prostate-cancer mortality at 11 years of follow-up. N Engl J Med. 2012 Mar 15;366(11):981-90. doi: 10.1056/NEJMoa1113135. PMID 22417251
- [Background] Andriole GL, Crawford ED, Grubb RL 3rd, Buys SS, Chia D, Church TR, Fouad MN, Gelmann EP, Kvale PA, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Clapp JD, Rathmell JM, Riley TL, Hayes RB, Kramer BS, Izmirlian G, Miller AB, Pinsky PF, Prorok PC, Gohagan JK, Berg CD; PLCO Project Team. Mortality results from a randomized prostate-cancer screening trial. N Engl J Med. 2009 Mar 26;360(13):1310-9. doi: 10.1056/NEJMoa0810696. Epub 2009 Mar 18. PMID 19297565
- See also: Cancer Incidence and Mortality Worldwide: IARC CancerBase — http://globocan.iarc.fr